CLINICAL TRIAL: NCT00394446
Title: Phase I Open Label, Dose Escalating, Multiple Dose Study to Determine the Safety, Tolerability, Maximum Tolerated Dose, and Pharmacokinetics of MPC-6827 Administered IV Weekly X 3, Repeated Every 28 Days, in Subjects With Refractory Solid Tumors.
Brief Title: Phase 1, Multiple Dose Study of MPC-6827 in Subjects With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Margaret Yu, MD / Director of Clinical Research, Myriad Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPC6827-04-001
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Refractory Solid Tumors
Keywords: Solid Tumors; Refractory; Brain
MeSH Terms: interventions — verubulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MPC-6827 — 2-hour intravenous infusion given once weekly for 3 consecutive weeks on a 28 day cycle

SUMMARY:
Phase 1, Multiple Dose Study of MPC-6827 in Subjects with Refractory Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or Metastatic Cancer
2. Measurable / Evaluable Disease
3. Karnofsky score greater than or equal to 70%
4. Adequate Hematology / Organ function
5. No Baseline peripheral or central neuropathy above grade 1

Exclusion Criteria:

1. Hypersensitivity to Cremophor EL
2. Pregnant or Lactating
3. Spinal Cord Compression
4. Pre-existing Dementia / Cognitive Disfunction
5. Require Neupogen or Neulasta to Maintain Neutrophil Count
6. Have Primary Brain Cancer
7. Have history of Ischemic Heart Disease
8. Have Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 year
Pharmacokinetics | 22 months

SECONDARY OUTCOMES:
Antitumor Activity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Yu, MD, Study Director — Myrexis Inc.
Locations (2):
- United States (2):
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah